CLINICAL TRIAL: NCT05525559
Title: A Phase I, Open-Label, Multi-Center Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of SHP2 Inhibitor ET0038 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: SHP2 Inhibitor ET0038 Monotherapy in Patients With Advanced Solid Tumors
Acronym: FIRST
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Etern BioPharma (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ET0038-101 US
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Oral capsules taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 21 days in duration with ET0038 administered, once daily (QD).
  Interventions: Drug: ET0038

INTERVENTIONS:
Drug: ET0038 — ET0038 for oral administration

SUMMARY:
This is a Phase I, open-label, multi-center, dose-finding study to assess the safety, pharmacokinetics, and preliminary efficacy of ET0038 in patients with advanced solid tumors. It is anticipated that approximately 34 subjects will be enrolled in the dose-escalation phase of the study. ET0038 will be administered orally once daily (QD) in 21-day treatment cycles.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1 study of oral ET0038 monotherapy in participants with advanced solid tumors. The study will include 2 components: 1) a Dose-Escalation Component for participants with advanced solid tumors and 2) a Dose-Expansion Component for participants with advanced solid tumors harboring certain specific mutations/rearrangements that result in hyperactivation of the RAS-MAPK pathway. Participants will be treated until disease progression per RECIST v1.1, unacceptable toxicity, or other criteria for withdrawal are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
2. Aged at least 18 years at the time of ICF signature.
3. Histological or cytological confirmation of a solid tumor and have progressed despite standard therapy(ies), or are intolerant to standard therapy (ies), or have a tumor for which no standard therapy(ies) exists. Locally recurrent disease must not be amenable to surgical resection or radiotherapy with curative intent (patients who are considered suitable for surgical or ablative techniques following down-staging with study treatment are not eligible).
4. Estimated life expectancy of minimum of 12 weeks.
5. Patient with solid tumors must have at least 1 lesion, not previously irradiated, that can be accurately measured at pre-dose as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with Computerised Tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at ICF signature.
7. Males and Females of child-bearing potential must agree to use effective contraception from the time ICF signature until 12 weeks after the last dose. Females of childbearing potential include those who are premenopausal and those who are 2 years postmenopausal. Pregnancy tests for female of child-bearing potential must have a negative serum pregnancy test at Screening.

Exclusion Criteria:

1. Primary central nervous system (CNS) tumor or uncontrolled CNS metastasis (severe clinical symptoms, bleeding, disease progression or steroid hormone use within 14 days before enrollment)..
2. As judged by the investigator, any evidence of significant ophthalmological abnormalities including but not limited to history or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO, retinal macular degeneration, uncontrolled glaucoma, cataract or marked decrease in visual acuity, symptomatic severe dry eye, conjunctivitis, or corneal ulcer.
3. Prior bone marrow or organ transplantation
4. Prior treatment with ET0038 or a SHP2 inhibitor.
5. Prior therapy with any investigational drugs or systemic anticancer treatment within 28 days (or a period of 5 'half-lives' of this investigational drugs or systemic anticancer treatment, whichever is the most appropriate and as judged by the investigator) at the time of ICF signature.
6. Radiotherapy with a wide field of radiation within 28 days, or radiotherapy with a limited field of radiation for palliation within 14 days at the time of ICF signature, or planning radical radiation therapy while participating in the study.
7. Prior major surgery (excluding placement of vascular access) within 28 days at the time of ICF signature, or planning for major surgery while participating in the study.
8. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE5.0) Grade 1 at the time of ICF signature.
9. Any uncontrolled active infection requiring parenteral administration of antibiotics, antivirals, or antifungals at the time of ICF signature and/or within one week of Cycle 1 Day 1 (C1D1).
10. Patient with a history of active pulmonary tuberculosis infection within 1 year prior to screening (as judged by investigator, active pulmonary tuberculosis infection more than 1 year and no evidence of active pulmonary tuberculosis at present will be considering eligible)
11. Patient with history or presence of interstitial lung disease or interstitial pneumonitis.
12. An active, or previously, autoimmune disease that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease,autoimmune thyroid disease, vasculitis, and psoriasis etc.) or high risk to such diseases.
13. Active infection including hepatitis B (Hepatitis B surface antigen [HBsAg] positive), and/or hepatitis C (HCV-RNA positive).
14. Active human immunodeficiency virus (HIV) infection (Patient with HIV positive and have well-controlled disease is exception).
15. Patient inability or unwillingness to comply with requirement for oral drug administration or presence of a gastro-intestinal condition, e.g., Refractory nausea and vomiting, inability to swallow the formulated product or previous significant bowel resection.
16. Have a history or present active bleeding disease within 6 months at the time of ICF signature.
17. History of COVID-19 infections, or COVID-19 nucleic acid test positive at the time of ICF signature and/or prior to the first dose of study treatment.
18. Pregnant or Breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) of ET0038 | Approximately 2 years
  MTD based on Number of participants with dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as any toxicity not attributable to the disease or disease-related processes under investigation, which occurs before the end of Cycle 1 (21 days as a cycle)
Recommended Phase 2 Dose (RP2D) | Approximately 2 years
  RP2D may be the same dose level or lower than the determined MTD.
Number of participants with adverse events | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments

SECONDARY OUTCOMES:
Area under the curve | Approximately 2 years
  Area under the plasma concentration time curve of ET0038
Cmax | Approximately 2 years
  Highest observed plasma concentration of ET0038
Tmax | Approximately 2 years
  Time of highest observed plasma concentration of ET0038
T1/2 | Approximately 2 years
  Half life of ET0038
Objective response rate | Approximately 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of response | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Disease Control Rate | Approximately 2 years
  DCR is defined as the percentage of patients who achieved remission (PR+CR) and stabilization (SD) after treatment in evaluable cases.
progression-free survival | Approximately 2 years
  PFS is defined as the time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
overall survival | Approximately 2 years
  OS is defined as the time between the beginning of randomization and the death of the patient from any cause

OTHER OUTCOMES:
Changes in phospho-ERK levels | Approximately 2 years
  Blood will be collected at pre-dose at screening and d on-treatment biopsy (between C2D1 and C3D1) to assess the extent of target engagement
NGS test of RTK/MAPK pathway genes | Approximately 2 years
  Next-generation sequencing (NGS) test will be performed with the tumor tissues or plasma ctDNA collected before ET0038 treatment, to detect gene alterations within the RTK/MAPK pathway. Detected gene alteration data (including but not limited to mutation, insertion, deletion, amplification, translocation…) will be further analyzed for correlation with the anti-tumor activity of ET0038.

CONTACTS AND LOCATIONS:
Locations (1):
- BUMC - Mary Crowley Cancer Research Centers (MCCRC), Dallas, Texas, United States